CLINICAL TRIAL: NCT01903889
Title: Promoting Constructive Male Engagement to Increase Use of Prevention of Mother to Child Transmission (PMTCT) Services
Brief Title: Male Engagement in PMTCT Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: Elizabeth Glaser Pediatric AIDS Foundation (Other); Mbarara University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 10385
Record Dates: First submitted 2013-07-17; First posted 2013-07-19 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: HIV
Keywords: AE adverse event; AIDS acquired immunodeficiency syndrome; ALT (SGPT) alanine aminotransferase; ART antiretroviral therapy; AST (SGOT) aspartate aminotransferase; DCF data collection forms; DMC Data Monitoring Committee; FDA (U.S.) Food and Drug Administration; GCP Good Clinical Practice guidelines; HB sAg Hepatitis B surface antigen; ICH International Conference of Harmonization; IND Investigational New Drug Application; IRB Institutional Review Board; IU International units; mg milligram(s); mm3 cubic millimeter(s); PCR polymerase chain reaction; SAE serious adverse event; µg microgram; ULN upper limit of the normal range; WB Western Blot; ANC Antenatal care; ARV Antiretroviral; C&T Care and treatment; CPR Contraceptive prevalence rate; DHS Demographic and Health Survey; EGPAF Elizabeth Glaser Pediatric AIDS Foundation; FP Family planning; HIV Human immunodeficiency virus; HTC HIV testing and counseling; IUCD Intrauterine contraceptive device; MCH Maternal/child health; PDA Personal digital assistant; PEPFAR President's Emergency Plan for AIDS Relief; PHSC Protection of Human Subjects Committee; PMTCT Prevention of maternal to child transmission; STAR-SW Strengthening TB and HIV/AIDS Response in the South Western Region of Uganda; STI Sexually transmitted infection; TM Technical monitor; USAID United States Agency for International Development; WHO World Health Organization
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases | interventions — Ambulatory Care Facilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinic based intervention (Active Comparator): basic intervention is introduced, whereby HIV/AIDS providers are trained on contraception for HIV-positive women. They are charged with counseling C&T clients on FP; offering condoms, pills and injectables; and referring clients for other FP methods
  Interventions: Other: clinic based intervention
- clinic and community based intervention (Experimental): The basic intervention is introduced along with an intervention for constructive male engagement in HIV and FP services. This includes training of C&T providers on gender-based influences on health behaviors; provision of couples' HIV testing and FP counseling services; and community-based education for men to promote gender equitable norms and male participation in health services.
  Interventions: Other: clinic and community based intervention

INTERVENTIONS:
Other: clinic based intervention — counseling C&T clients on FP; offering condoms, pills and injectables; and referring clients for other FP methods
  Arms: Clinic based intervention
Other: clinic and community based intervention — basic intervention is introduced along with an intervention for constructive male engagement in HIV and FP services
  Arms: clinic and community based intervention

SUMMARY:
The study employs a quasi-experimental design in 8 public health centers in southwest Uganda offering care and treatment (C&T) services. In 4 health centers, a basic intervention is introduced, whereby HIV/AIDS providers are trained on contraception for HIV-positive women. They are charged with counseling C&T clients on FP; offering condoms, pills and injectables; and referring clients for other FP methods. In the other 4 health centers, the basic intervention is introduced along with an intervention for constructive male engagement in HIV and FP services. This includes training of C&T providers on gender-based influences on health behaviors; provision of couples' HIV testing and FP counseling services; and community-based education for men to promote gender equitable norms and male participation in health services.

DETAILED DESCRIPTION:
This study will be conducted in Kabale District, Uganda, a rural district where prevention of mother to child transmission (PMTCT) and care and treatment (C&T) services are offered in eight public sector health facilities. The primary aim of this study is to test an intervention for increasing use of the full spectrum of PMTCT services, including family planning (FP), through enhanced constructive male involvement in reproductive health decision making. This aim will be accomplished by conducting a cluster randomized trial, whereby a "constructive male engagement" intervention package will be introduced in four randomly selected health centers and surrounding communities; the other four sites will serve as comparisons. Pre- and post-intervention cross sectional surveys will be conducted with male and female C&T clients to assess intervention effectiveness, measured in terms of dual method use. In addition to the male engagement intervention, reinforcements will be introduced in all eight participating facilities to enhance providers' capacity to serve the FP needs of C&T clients. We hypothesize that the percentage of clients reporting dual method use will increase slightly in all facilities as a result of this "HIV-FP integration intervention." To measure the independent effect of the reinforcements, the study will compare contraceptive knowledge, attitudes, and behaviors of clients measured pre- and post-intervention in the comparison sites only, in the absence of the male engagement intervention. We further hypothesize that improvements will be incrementally greater in the four facilities exposed to the additional constructive male engagement intervention.

The study will include additional data collection and analyses to support secondary objectives.

1. Services statistics will be tracked to assess changes in uptake and continuation of PMTCT services.
2. The study will include a qualitative component to investigate condom use behaviors. Based on other investigations, it is anticipated that rates of self-reported condom use among C&T clients will be high. To examine those behaviors more closely and to circumvent courtesy bias often associated with quantitative surveys, the study will conduct individual in-depth interviews with a subset of female and male C&T clients reporting consistent condom use.
3. The constructive male engagement intervention will comprise both community- and clinic-based components. To assess the effectiveness of the community-based men's workshops, the study will assess changes in knowledge, attitudes, and behaviors among men exposed to the community-based intervention by surveying them before and 4 months after community-level training is held. Interviews will assess knowledge and attitudes related to FP and HIV services (PMTCT in particular), with particular focus on gender norms supporting constructive male involvement. Interviews will also examine clients' recollection of services and messages received in the health center, along with their direct and indirect exposure to the community-based men's workshops.
4. The effectiveness of the intervention components aimed at reinforcing the capacity of clinic-based providers to serve the family planning needs of HIV-positive individuals and to engage male partners constructively in FP decision making will be assessed in terms of its impact on C&T clients. Specifically, interviews with C&T clients will include questions about messages communicated by providers and service delivery practices reflecting successful implementation of the intervention components.
5. Finally, the study will examine the resource requirements for adding each the interventions (reinforcement of FP and male involvement) into C&T services. Based on costs of the piloted interventions, the study will arrive at an estimate of the cost of implementing these interventions at scale under the direction of the district management team.

ELIGIBILITY:
Inclusion Criteria:

female participants

* attending pre-ART and ART services;
* non-pregnant women;
* age 18 to 45;
* sexually active with any type of partner within the past 3 months.

male participants

* attending pre-ART and ART services;
* age 18 to 60;
* sexually active within the past 3 months with partner, either co-habiting partner or steady, with partner aged 18 to 45 and is not pregnant.

Exclusion Criteria:

* For the post-intervention interviews, clients who initiated Care & Treatment services in one of the intervention facilities less than 3 months prior will be excluded given insufficient exposure to the intervention.
* Clients unable to speak Runyankole, the dominant language in the region, will also be excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3806 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
To assess the effectiveness of an intervention aimed at constructively engaging men in FP decision making | 12 months
  Dual method use among couples with at least one partner using C&T services

SECONDARY OUTCOMES:
To measure changes over time in uptake of Prong 3 PMTCT services, comparing facilities that are and are not exposed to the constructive male engagement intervention | 6 months
  Number of new ANC clients
To assess the effect of reinforcements introduced to enhance C&T providers' capacity to serve the FP needs of HIV-positive clients, as reflected in C&T clients' knowledge, attitudes, and behaviors related to FP. | 12 months
  Dual method use among couples with at least one partner using C&T services 2) Knowledge and attitudes related to FP
To explore condom use dynamics and the factors favoring and discouraging consistent use by cohabiting couples | 1 month
  1) Consistency of condom use 2) Factors encouraging and impeding consistent condom use
To evaluate men's knowledge and attitudes related to gender norms and FP and HIV services before and after participation in a 10-week community education and mobilization program. | 10 months
  1) Perspectives on acceptable gender norms 2) Knowledge, attitudes, and behaviors related to use of family planning and HIV services.
To document the technical, human, and material resources required to implement the study interventions and to estimate the financial cost of implementation at scale. | 12 months
  Cost of implementing HIV-FP integration intervention and male engagement intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Hoke, Ph.D., MPH, Principal Investigator — FHI 360
Locations (7):
- Uganda (7):
  - Bukinda Health Center, Kabale
  - Kamkira Health Center, Kabale
  - Kamwezi Health Center, Kabale
  - Maziba Health Center, Kabale
  - Mparo Health Center, Kabale
  - Muko Health Center, Kabale
  - Rubaya Health Center, Kabale